CLINICAL TRIAL: NCT02463877
Title: A Minimally-invasive Approach to Cytoreduction and HIPEC for Peritoneal Surface Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dr. Kaitlyn J Kelly, Assistant Clinical Professor of Surgery, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minimally-Invasive
Record Dates: First submitted 2015-04-20; First posted 2015-06-04 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Minimally-Invasive Procedure (Experimental): single-arm study of laparoscopic cytoreduction and HIPEC
  Interventions: Procedure: Minimally-Invasive Procedure

INTERVENTIONS:
Procedure: Minimally-Invasive Procedure — Laparoscopy

SUMMARY:
The purpose of this study is to determine the feasibility of surgical techniques involving minimal entry into the living body approach for tumor reduction and treatment in which highly concentrated anticancer drugs are put directly into the abdomen through a tubes (HIPEC), and to determine if this approach may improve short-term postoperative outcomes, including the development of complications related to surgery within the first 30 days after surgery.

Participation in this study is entirely voluntary. Approximately 30 subjects will take part in this single-center study and all will be enrolled at University of California San Diego.

DETAILED DESCRIPTION:
Potential patients will be prospectively identified prior to the time of operation based on the inclusion/exclusion criteria . Those who meet the eligibility criteria and sign consent will undergo laparoscopy. During laparoscopy, the peritoneal cancer index (PCI) will be determined for all patients. The PCI is a scoring system that was developed to standardize the assessment of disease burden. PCI is determined by assigning a Lesion size score (LSS) to each of the 13 peritoneal regions and then summing the scores (defined further below). Those with a PCI of ≤10 will continue with laparoscopic cytoreduction and HIPEC. Patients with a PCI of >10 will have an open cytoreduction and HIPEC. The Investigators plan to enroll 30 patients, though the investigators estimate 18 will ultimately undergo laparoscopic cytoreduction and HIPEC.

Trial Design:

* Stage 1 will enroll 9 patients, and if 2 or less patients experience postoperative complications within 30 days of HIPEC the investigators will proceed to stage 2. If 3 or more patients experience postoperative complications the investigators will terminate the trial early secondary to futility.
* Stage 2 will enroll 9 additional patients, and if the investigators have 4 or less patients with postoperative complications out of the total 18 patients the investigators will reject the null hypothesis.

Visit 1- screening

* History and physical examination
* Routine blood tests standard for monitoring of patient's disease include a complete blood count, kidney and liver chemistries, and tumor markers (CEA and carbohydrate antigen 19-9 (CA19-9)) if not already performed;
* Imaging tests per standard of care (chest x-ray, CT scan; PET Scan); possibly laparoscopy or colonoscopy (both scan patients abdomen area); if not performed prior to consultation at University of California, San Diego (UCSD)
* Electrocardiogram (ECG); thallium heart scan or echocardiogram if history of cardiac disease (prior Myocardial Infarction, Congestive Heart Failure, angina, cardiomyopathy, vascular dysfunction and arrhythmia)

Visit 2 - operation/ surgery

* Physical exam and updated medical history
* Routine blood tests
* Laparoscopic exploration prior to cytoreduction, will be performed, per local standard of care for assessment of PCI.
* HIPEC will be administered per local standard of care..
* A greater omentectomy will be performed routinely in all cases as is done in open cytoreduction. Greater and lesser omentectomy, omental bursectomy, splenectomy, left and right upper quadrant and pelvic peritonectomy, cholecystectomy, total abdominal hysterectomy, low anterior resection and/or gastrectomy will be performed at the surgeon's discretion based on volume and distribution of peritoneal surface malignancy with the aim of achieving complete resection of all grossly apparent disease.
* Peritonectomy and organ resection will be performed to achieve optimal cytoreduction (defined as removal of all gross disease or cytoreduction to gross deposits less than 2.5 mm in thickness).
* If it is determined that optimal cytoreduction cannot be achieved with minimally-invasive techniques, the procedure will be converted to an open operation.
* Laparotomy -In cases where minimally-invasive optimal cytoreduction is achieved, a small (4 to 6 cm) laparotomy incision will be made when necessary for organ extraction and a wound protector will be used. The mini-laparotomy incision will be utilized for insertion of HIPEC catheters.
* Temporary skin closure will be performed at all port sites and incisions for closed-HIPEC. Bowel anastomoses and fascial closure of port sites ≥ 1 cm and of mini-laparotomy incisions will be performed after completion of HIPEC.
* Completeness of cytoreduction will be estimated and recorded using the system shown below. Intra-peritoneal tubes and drains will be placed at the surgeon's discretion and the incision closed in the usual fashion.
* After the procedure, the patient will stay in the intensive care unit (ICU) for about 24-48 hours. For at least 4 hours after the procedure the patient will be asked to stay in bed. The patient will then stay in the hospital for approximately 3-5 days after the procedure. This is part of the standard of care.

Surgery must start within 8 weeks from time of screening. Surgery must be performed by a surgeon experienced in cytoreductive and HIPEC surgery who has met the credentialing requirements of the study.

Pre-perfusion protocol and perfusion circuit set-up and priming:

At the conclusion of cytoreductive surgery, hemodynamic stability of the patient will be assured and bleeding points controlled per standard of practice. Systemic body temperature will be monitored. The perfusion system will be assembled per the operator's manual utilizing sterile technique. The perfusion circuit priming will be with a balanced electrolyte solution; 1.5% Delflex Peritoneal Dialysis (DPD) solution is preferred. In the absence of ascites, approximately 3-4 Liters of perfusate is required for the circuit and priming in an average 70-kg adult. A general guideline is 1.5-2.0 L/m2 perfusate. The perfusate will be primed, heated to target temperature at the discretion of the operating surgeon and re-circulated.

After a patient receives their cytoreductive surgery and HIPEC whether by minimal invasive or open approach, the biohazardous fluid is collected in the chemotherapy waste containers for disposal.

Placement of inflow and outflow catheters and temperature probes Peritoneal perfusion catheters and temperature probes will be placed by the operating surgeon in accordance with standards of practice. Inflow catheter positioning in the sub-diaphragmatic region of the peritoneal cavity is preferred. Outflow catheter positioning in the pelvis is preferred. This protocol allows for open delivery of heated chemotherapy at surgeon discretion. Timing of intestinal reconstruction and formation of stomas will be at surgeon discretion. Sterile pump lines from the perfusion system will be delivered to the sterile field and the lines will be filled with perfusate to prevent airlocks. The inflow and outflow tubing will be connected and the pre-heated perfusate will be allowed to fill the peritoneal cavity. Usually ~3 liters of solution is required to distend the cavity and achieve desired flow rates.

Recommended anesthetic management and intra-operative physiological monitoring during HIPEC An epidural catheter may be placed at the discretion of the operating team (anesthesiologist and surgeon). Broad-spectrum antimicrobial prophylaxis is recommended prior to surgical incision (specific antibiotic at the discretion of the operating surgeon). Radial arterial cannulation may be established for arterial-line blood pressure monitoring. A triple lumen central venous catheter may be placed at the anesthesiologist's discretion. A nasogastric tude is typically placed to decompress the stomach. A transurethral catheter is placed in the bladder. During cytoreductive surgery, careful attention to end tidal carbon dioxide, oxygen saturation and peak airway pressures is made during diaphragmatic stripping assessing for signs of pneumothorax. The patient's core body temperature may be reduced to 35 degrees Celsius (95 °F) prior to commencing hyperthermic intraperitoneal chemotherapy. At the start of the hyperthermic chemotherapeutic infusion, the Bair Hugger may be set to blow ambient air flow over the patient. Adequate intravenous fluid hydration with crystalloid and/or colloid prior to initiation of the hyperthermic chemotherapeutic perfusion is important, as systemic vasodilatation occurs during the perfusion. Urinary output during HIPEC should be maintained at 0.5-1.0 ml/kg/hr. Clotting time and INR, serum electrolytes, blood gases, and vital signs are monitored throughout the procedure. Standards of anesthetic practice interventions should occur when clinically appropriate. Fresh frozen plasma is utilized to maintain INR ≤ 1.5 as appropriate

* Heated intraoperative intraperitoneal chemotherapy will be delivered as above. At the completion of the perfusion, the abdomen will be re-explored, residual fluid aspirated, bleeding points controlled and reconstructive operation completed if not already done prior to HIPEC (anastomosis with or without diverting stoma).
* Mitomycin C will be the agent administered for patients with primary appendiceal and colorectal cancers at a dose of 30 mg/kg. For rare cases of primary peritoneal mesothelioma or ovarian primary tumors, Cisplatin ( 50 mg/m2) or Doxorubicin (15 mg/m2) may be used. This is the current standard of care and is not specific to this trial protocol.

Follow up visits- A follow up visit after 2 weeks and 6 weeks of the surgery for physical exam and updated medical history.

Then every 3 months (+/- 2 weeks) for the first three year, every 6 months for the next 2 years, and yearly thereafter if no evidence of recurrence. The patient will need the following tests and procedures during routine follow-up visits. These are part of regular cancer surveillance and care and are not specific to this study.

Physical exam and updated medical history; Pain assessment; Routine blood tests and study blood tests; Cross-sectional imaging with CT scan or MRI per standard of care

If patients develop symptoms or exam findings warranting cross-sectional imaging at different time points, imaging will be performed as needed.

Data collected includes demographics (age, gender), past medical history, past surgical history, weight, body mass index, body surface area, ICU length of stay, hospital length of stay, IV narcotic requirements, time to return of bowel function, need for and duration of Nasogastric tube (NGT) decompression, diagnosis, surgical procedures performed, HIPEC agents administered, operative time, estimated blood loss, and postoperative complications will be recorded. Postoperative complications are defined according to the validated classification system proposed by Clavien and colleagues.8 Briefly, a complication is defined as any deviation from the normal postoperative course. Complications are classified according to the involved organ system and are graded according to the therapy required to treat the complication. Grade I complications are deviations from the expected / normal course, but do not require pharmacologic, surgical, endoscopic, or radiological intervention for treatment. Grade II complications require pharmacologic intervention, including blood transfusion and total parenteral nutrition. Grade III complications require surgical, endoscopic, or radiological intervention. Grade IV complications are defined as life-threatening events requiring intensive care for management. Grade V complication is defined as death.

For assessment of oncologic outcomes, patients will be followed with clinic visits every 3 months for the first year, then every 6 months for the next 2 years, and yearly thereafter if no evidence of recurrence. For patients with recurrent disease, data will be collected on: site of recurrence, date of recurrence, disease status (no evidence of disease, alive with disease, died from disease, or died of unknown cause), and length of follow-up will be recorded. This data will be extracted from the patients' medical records for 5 years from the time of initial Institutional Review Board (IRB) approval.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 18 years old
2. Capable of providing informed consent.
3. Histologically confirmed peritoneal carcinomatosis from appendiceal, colorectal, ovarian, or primary mesothelioma, with no systemic metastases.
4. Evidence of low-volume peritoneal disease defined by a PCI < 10 based on cross-sectional imaging / and / or diagnostic laparoscopy findings.
5. Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status of 0-2.
6. Patients who are medically fit for surgery defined as the following:

   * No parenchymal hepatic metastases
   * No evidence of clinical (jaundice), biochemical (abnormally elevated serum bilirubin and/or alkaline phosphatase) or radiological (ultrasound, CT, or MR) biliary obstruction
   * No cross sectional imaging findings indicative of multi-segmental (>1 site) small bowel obstruction, or small bowel loops matted together, or gross disease of the small bowel mesentery characterized by distortion, thickening or loss of mesenteric vascular clarity
   * No clinical or radiological evidence of hematogenous or distant nodal (retroperitoneal, pelvic, mediastinal, peri-portal or peri-aortic) metastasis
   * Absolute neutrophil count (ANC) > 1200/mm3, white blood cell count (WBC) > 4000/mm3 and platelet count > 150,000/mm3
   * An international normalized ratio (INR) ≤ 1.5 (patients who are therapeutically anticoagulated for unrelated medical conditions such as atrial fibrillation and whose antithrombotic treatment can be withheld for operation will be eligible).
   * Adequate hepatic function must be met as evidenced by total serum bilirubin ≤ 1.5 mg/dl (patients with total bilirubin > 1.5 mg/dL eligible only with Gilbert's syndrome);
   * Alkaline phosphatase < 2.5 times the upper limit of normal; and/or
   * Aspartate transaminase (AST) < 1.5 times upper limit of normal (alkaline phosphatase and AST cannot both exceed the upper limit of normal)
   * Serum renal functional parameters, blood urea nitrogen (BUN) and creatinine are within normal limits
   * Satisfactory cardiopulmonary function (no history of severe congestive heart failure or severe pulmonary disease, as indicated by clinically acceptable risks to undergo major abdominal - cytoreductive surgery).
   * No clinical history of acute myocardial infarction within six months of registration.
   * Patients who are status post revascularization procedures with satisfactory cardiac function are eligible.
   * No significant history of a medical problem or co-morbidity that would preclude the patient from undergoing a major abdominal operation such as a history of severe congestive heart failure or active ischemic heart disease.
7. No concurrent second malignancy requiring systemic therapy.
8. No psychiatric or addictive disorders or other conditions that would preclude the patient from meeting the study requirements.

Exclusion Criteria:

1. Peritoneal carcinomatosis index (PCI) > 10
2. Systemic (extraperitoneal) disease, pregnant, incarcerated.
3. Pregnant and lactating women. Women of reproductive age must be willing to use contraception during study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative complications | within 30 days of surgery
  Rate of postoperative complications within 30 days of surgery: this will be expressed as simple ratio with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn Kelly, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with Genelux Corporation

REFERENCES:
- [Derived] Cho CY, Veerapong J, Baumgartner JM, Murphy JD, Lowy AM, Kelly KJ. Laparoscopic cytoreductive surgery and hyperthermic intraperitoneal chemotherapy: a prospective clinical trial and comparative analysis. Surg Endosc. 2023 Jul;37(7):5644-5651. doi: 10.1007/s00464-022-09589-w. Epub 2022 Dec 7. PMID 36477643